CLINICAL TRIAL: NCT04443465
Title: Physical Effects and Emotional Experiences of Intra-operative Neuro-monitoring (IONM)
Brief Title: Patient Experiences of IONM and Outcomes
Acronym: IONM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 239002
Record Dates: First submitted 2018-10-10; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-03

CONDITIONS: Intraoperative Neurophysiological Monitoring; Complication; Intraoperative Complications; Postoperative Complications
MeSH Terms: conditions — Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Resection of brain tumours forms a large proportion of work in brain surgery. One important aspect is to minimize damage to normal brain structures during this process. This improves patient outcomes and reduces complications. To identify normal brain structures from the abnormal tumours, the brain surgeons use a 'guidance' technique called intraoperative neuro-monitoring (IONM).

IONM uses various electrodes to observe spontaneous electrical activity of the brain or its reaction to a stimulus such as muscle contraction, light or sound. It is now becoming common practice for neurosurgeons to use this tool during brain and spinal surgery to provide a real-time feedback under anaesthesia to help them minimise injury to important and normal brain and spine structures.

IONM interpretation needs fulfilment of multiple preconditions and major modifications to the anaesthetic to reduce its inaccuracies. This invites added risks and complications such as awareness, convulsions and heart problems under anaesthesia. A team approach between the surgeon, anaesthetist and neurophysiologist (IONM specialist) is also crucial to obtain meaningful results. Therefore, the usefulness of this technique is still not perfect.

Although, benefits of IONM are obvious, information on associated complications and patient experience are not commonly found in the literature. Information on other effects such as hormonal balance and tumour recurrence are also scarce. In general, these aspects have little scientific exploration.

There are anecdotal reports of recurrent seizures during IONM leading to serious heart problems, teeth and tongue damage due to grinding and postoperative calf muscle injury necessitating further surgery to save limbs. Neither of these is in the literature including unorthodox treatments such as the use of cold saline to control IONM triggered fits.

This study is designed to observe complications and outcome and explore patient experiences following IONM in an observational capacity not interfering with the clinical management or treatment of these patients. The investigators intend to interview the participants after surgery, at a convenient time before leaving hospital to understand their views and experiences during and after surgery and their general progress in the following one year.

DETAILED DESCRIPTION:
INTRODUCTION Intraoperative neuro-monitoring (IONM) is a 'SAT NAV' used by neurosurgeons to prevent injury to normal structures during brain and spinal surgery under anaesthesia. It involves the use of surface and implanted electrodes to observe spontaneous electrical activity of the brain or evoked responses to an electrical stimulus (motor, visual or auditory). This requires major modifications to the anaesthetic that provides lighter planes of anaesthesia with no muscle relaxation inviting added risks and complications such as awareness, seizures and cardiac events.

This cohort study over a period of one year will include a qualitative enquiry of patient experience and a quantitative evaluation of the immediate postoperative course and complications at 28 days and 1 year. It will explore the relatively unknown area of emotional experiences of participants under anaesthesia who undergo various types of neuro stimulation and related post-operative sequelae. The results are expected to assist improve patient experiences and outcomes.

BACKGROUND AND RATIONALE Resections of brain tumours constitute a significant proportion of work in neurosurgery. One important aspect is minimizing injury to normal neural structures during this process to improve outcomes of such operations and reduce complications. This involves intraoperative neuro-monitoring (IONM).

IONM uses surface and implanted electrodes to observe spontaneous electrical activity of the brain or evoked response to a motor, visual or auditory stimulus. It is now becoming common practice for neurosurgeons to use this tool during brain and spinal surgery to provide a real-time feedback under anaesthesia to help them minimise injury to critical and normal neural structures by 'mapping' normal from abnormal areas of the brain.

IONM interpretation needs fulfilment of multiple preconditions and major modifications to the anaesthetic to reduce its inaccuracies. This invites added risks and complications such as awareness, seizures and cardiac events. A team approach is also crucial to obtain meaningful results. Therefore, the utility of this technique is still evolving based on personal experiences and perceptions and the understanding between the surgeons, anaesthetists and neurophysiologists.

Although, benefits of IONM are obvious, data on associated post-operative morbidity and patient experience and complications are scarce. The data is also scarce on tumour recurrence or tumour behaviour following IONM guided neurosurgery. More precise excision may reduce tumour recurrence. On the other hand IONM related electrical stimulation may impose humoral effects on tumour behaviour. These aspects have little scientific exploration.

There are anecdotal reports of recurrent seizures during IONM leading to cardiac events such as asystole, teeth grinding and damage and tongue injury in the absence of a 'bite block' and postoperative calf muscle necrosis necessitating fasciotomies. Neither of these is in the literature including the unorthodox effective treatments used such as pouring 'cold' saline on the surface of the brain to control seizures.

The study will take place in a major neurosurgical centre in the UK that uses IONM. Therefore, the study population is vast for appropriate sampling and recruitment.

STUDY DESIGN This is an observational cohort study based on data retrieved from clinical notes and direct patient interview in hospital. The qualitative enquiry will address emotional aspects and the process experience. The quantitative survey will investigate morbidity (post-operative recovery, complications) and outcomes including mortality at 28 days and 1-year follow-up.

The eligible patients will be identified by the published elective neurosurgery lists and approached for informed consent before surgery at the time of preoperative assessment.

The anaesthetist or the surgeon directly involved with his/her clinical care will first approach the patient and subsequently introduced to the medical student for post-operative data collection. Their demographic data, disease data, and neurological assessment scores will be obtained from medical records. Direct patient interviews will be carried out by the investigators postoperatively, using a structured open questionnaire format. This activity will merge with the postoperative clinical rounds where possible.

All patients undergoing elective neurosurgery guided by IONM will be eligible for the study and recruited with informed consent. The exclusion criteria shall be aged less than 10 years, lack of informed consent and who are unable to communicate verbally.

A convenient sample of 50 is a realistic number of patients who can be recruited within a 3-month period at this centre. However, the qualitative enquiry may be stopped at an earlier time if the data collected is felt to be at the saturation point by the investigators. The participants shall be followed up at 28 days and 1-year post surgery.

Continuous data will be described and analysed based on their distribution, be it parametric or non-parametric. Dichotomous data will be described as number of patients/episodes and percentage.The patient experiences reported will be subjected to a thematic analysis following the principles of qualitative research grounded theory.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 10 and above undergoing elective neurosurgery guided by IONM will be recruited with informed consent.

Exclusion Criteria:

* Lack of informed consent and who are unable to communicate verbally.-

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children aged 10 and above undergoing brain or spinal surgery with intra operative neurophysiological monitoring with intravenous anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Experiences of participants who undergo intra-operative neurophysiological monitoring under anaesthesia | 2 years
  A qualitative study of patient experiences by thematic analysis

SECONDARY OUTCOMES:
IONM related postoperative sequel during post surgical recovery in hospital | 2 years
  Perioperative adverse events description
Mortality at 28 day and 1 year follow up | 2 years
  Mortality rates at 28 days and 1 year
Morbidity at 28 days and 1 year follow up | 2 years
  Residual weaknesses and disability

CONTACTS AND LOCATIONS:
Overall Officials: Chulananda Goonasekera, PhD, Principal Investigator — Kings College Hospital NHS Trust, London
Locations (1):
- Kings College Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised qualitative and quantitative data

REFERENCES:
- [Background] Stecker MM. A review of intraoperative monitoring for spinal surgery. Surg Neurol Int. 2012;3(Suppl 3):S174-87. doi: 10.4103/2152-7806.98579. Epub 2012 Jul 17. PMID 22905324
- [Background] Jameson LC, Sloan TB. Monitoring of the brain and spinal cord. Anesthesiol Clin. 2006 Dec;24(4):777-91. doi: 10.1016/j.atc.2006.08.002. PMID 17342964
- [Background] Arnold PM. Use of intraoperative monitoring in children. J Neurosurg Pediatr. 2014 Jun;13(6):589. doi: 10.3171/2013.9.PEDS13439. Epub 2014 Apr 4. No abstract available. PMID 24702618
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Result] Jameson LC, Janik DJ, Sloan TB. Electrophysiologic monitoring in neurosurgery. Anesthesiol Clin. 2007 Sep;25(3):605-30, x. doi: 10.1016/j.anclin.2007.05.004. PMID 17884710
- [Result] Soghomonyan S, Moran KR, Sandhu GS, Bergese SD. Anesthesia and evoked responses in neurosurgery. Front Pharmacol. 2014 Apr 14;5:74. doi: 10.3389/fphar.2014.00074. eCollection 2014. No abstract available. PMID 24782777
- [Result] Cabraja M, Stockhammer F, Mularski S, Suess O, Kombos T, Vajkoczy P. Neurophysiological intraoperative monitoring in neurosurgery: aid or handicap? An international survey. Neurosurg Focus. 2009 Oct;27(4):E2. doi: 10.3171/2009.7.FOCUS0969. PMID 19795951

DOCUMENTS (1):
  • Informed Consent Form (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04443465/ICF_000.pdf